CLINICAL TRIAL: NCT05936710
Title: Improved Hemodynamic Tolerance of Intermittent Hemodialysis Sessions in Intensive Care Unite (ICU) Using Citrate- vs Acetate-based Dialysate
Brief Title: Improved Hemodynamic Tolerance of Intermittent Hemodialysis Sessions in Intensive Care Unite Using Citrate- vs Acetate-based Dialysate
Acronym: HEMODIACIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Bethune (Network)
Collaborators: CHU de Lille (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-01
Record Dates: First submitted 2023-05-19; First posted 2023-07-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Intradialytic Hypotension
Keywords: citrate based dialysate; acetate based dialysate; hypotension; hemodynamic tolerance
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Using acetate-based dialysate
  Interventions: Device: ACETATE based dialysate
- Experimental group (Experimental): Using citrate-based dialysate
  Interventions: Device: CITRATE based dialysate

INTERVENTIONS:
Device: ACETATE based dialysate — Intermittent hemodialysis with an acetate based dialysate.
  Arms: Control group
Device: CITRATE based dialysate — Intermittent hemodialysis with an citrate based dialysate.
  Arms: Experimental group

SUMMARY:
During intermittent hemodialysis (IHD), the occurrence of intradialytic hemodynamic instability (IHI) is frequent in ICU and impacted morbidity and mortality. Bicarbonate dialysate buffer improves hemodynamic tolerance compared to acetate dialysate buffer. However, bicarbonate dialysate buffer still contains a lower concentration of acetate, which could contribute to hemodynamic instability. Recently, citrate-based dialysate in bicarbonate hemodialysis instead of acetate have been proposed. They have the appropriate authorizations for routine use. The aim of this study is to compare acetate- vs citrate-based dialysate in terms of hemodynamic tolerance and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years old
* Patient hospitalized in an intensive care unit
* Patient with acute renal failure defined by a KDIGO stage ≥ 1 and suspected non-obstructive
* Patient at risk of per dialytic hypotension (capillary refill time ≥ 3 seconds and/or cardiovascular SOFA ≥ 1 and/or lactatemia > 2mmol/L)
* Indication for Extra Renal Replacement Therapy with IHD.

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Known chronic renal insufficiency of any stage
* Cardio-renal and hepato renal syndrome
* Unstable hemodynamic state: refractory shock
* Patient included in another interventional study likely to modify the hemodynamic state
* Patient deprived of liberty
* Patient under guardianship or curatorship
* Patient not affiliated to a social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
To show that the use of a citrate-based dialysate decreases the occurrence of intradialytic hypotension in the ICU compared with an acetate-based dialysate (The rate of sessions with occurence of at least one hemodynamic instability (IHI)). | day 28
  The rate of sessions with occurence of at least one IHI.

SECONDARY OUTCOMES:
Compare between the two groups (acetate- vs citrate-based dialysate) the mortality at day 28 and in ICU; | day 28
  Mortality at day 28 and in ICU;
Compare between the two groups (acetate- vs citrate-based dialysate) the length of stay in Intensive Care Unit. | day 28
  Length of stay in Intensive Care Unit
Compare between the two groups (acetate- vs citrate-based dialysate) the Length of stay in hospital. | day 28
  Length of stay in hospital;
Compare between the two groups (acetate- vs citrate-based dialysate) the Number of days without dialysis in Intensive Care Unit. | day 28
  Number of days without dialysis in Intensive Care Unit
Compare between the two groups (acetate- vs citrate-based dialysate) the dialysis dependency at discharge from ICU and hospital. | day 28
  Dialysis dependency at discharge from ICU and hospital.
Compare between the two groups (acetate- vs citrate-based dialysate) the time to recovery of diuresis > 0.5ml/kg/h. | day 28
  Time to recovery of diuresis > 0.5ml/kg/h
Compare between the two groups (acetate- vs citrate-based dialysate) the change in SOFA score between D0 and D7. | day 28
  Change in SOFA score between D0 and D7
Compare between the two groups (acetate- vs citrate-based dialysate) the number of days without catecholamine. | day 28
  Number of days without catecholamine
Compare between the two groups (acetate- vs citrate-based dialysate) the number of days without mechanical ventilation. | day 28
  Number of days without mechanical ventilation.
Compare between the two groups (acetate- vs citrate-based dialysate) the ratio of Kt/V (achieved/prescribed). | day 28
  The ratio of Kt/V (achieved/prescribed)
Compare between the two groups (acetate- vs citrate-based dialysate) session duration ratio (duration achieved/prescribed). | day 28
  Difference between session duration achieved and prescribed
Compare between the two groups (acetate- vs citrate-based dialysate) UF ratio (UF prescribed/realized) | day 28
  UF ratio (UF prescribed/realized)
Compare between the two groups (acetate- vs citrate-based dialysate) urea reduction rate (pre-dialysis urea - post-dialysis urea/pre-dialysis urea) | day 28
  Urea reduction rate (pre-dialysis urea - post-dialysis urea/pre-dialysis urea)
Compare between the two groups (acetate- vs citrate-based dialysate) average, maximum and end-of-session blood and dialysate flow rates. | day 28
  Average, maximum and end-of-session blood and dialysate flow rates.
Compare between the two groups (acetate- vs citrate-based dialysate) the pre-post dialysis variation in creatinine levels. | day 28
  The pre-post dialysis variation in creatinine levels
Compare between the two groups (acetate- vs citrate-based dialysate) the pre-post dialysis variation of pH and bicarbonate level. | day 28
  The pre-post dialysis variation of pH and bicarbonate level
Compare between the two groups (acetate- vs citrate-based dialysate) the pre-post dialysis variation in kalemia. | day 28
  The pre-post dialysis variation in kalemia
Compare between the two groups (acetate- vs citrate-based dialysate) the pre-post dialysis the rate variation of sodium, magnesium and calcium. | day 28
  The pre-post dialysis rate variation of sodium, magnesium and calcium
Compare between the two groups (acetate- vs citrate-based dialysate) the rate of calcium supplemented between two IHD sessions. | day 28
  The rate of calcium supplemented between two IHD sessions.
Evaluate the hemodynamic tolerance | Each dialysis until day 28
  according to the randomization groups : the response to the passive leg raising, respiratory variation of the inferior vena cava etc...

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Centre Hospitalier Béthune, Béthune
  - CHU, Caen
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - CHRU Nancy, Nancy